CLINICAL TRIAL: NCT06980376
Title: Effects of Milk Free From A1-Type β-Casein on Inflammation, Gastrointestinal Tolerance, and Pregnancy Outcomes: A Multi-Centre, Randomised, Open-Label, Prospective Study
Brief Title: Milk Free From A1-Type β-Casein on Inflammation, Gastrointestinal Tolerance, and Pregnancy Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Collaborators: Edanz Inc (Unknown); Cyanth (Wuxi) Health Technology Co. Ltd. (Unknown); Affilicated Hospital of Jiangnan University (Unknown); Guangzhou Trials Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A2MC-G2411-73081
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Healthy Pregnant Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a2 UHT Milk (Active Comparator): containing A2 type β-casein only (A1PF)
  Interventions: Other: a2 UHT milk
- Conventional UHT milk (Placebo Comparator): containing both A1 and A2 type β-caseins (CON)
  Interventions: Other: Conventional UHT Milk

INTERVENTIONS:
Other: a2 UHT milk — Pregnant women in this arm will drink a2 UHT Milk twice a day, 200ml each time, until study completion. Their infants will be fed with the mother's breastmilk exclusively.
  Arms: a2 UHT Milk
Other: Conventional UHT Milk — Pregnant women in this arm will drink conventional UHT Milk twice a day, 200ml each time, until study completion. Their infants will be fed with the mother's breastmilk exclusively.
  Arms: Conventional UHT milk

SUMMARY:
The aim of the study is to compare the effects of conventional Ultra High Temperature (UHT) milk containing both A1 and A2 type β-caseins (CON) with a2 UHT Milk containing A2 type β-casein only (A1PF) on inflammation, tolerance, and GI symptoms in pregnant women as well as infants' birth outcomes from 12 weeks' gestation up to 40 days post-birth.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years of age
* Recruited at <12 weeks of gestation
* Intention to deliver at study site hospital
* Singleton pregnancy
* Able and willing to consume milk during pregnancy
* Agree not to participate in another interventional clinical study during the present study

Exclusion Criteria:

* Body mass index ≥ 35 at enrolment
* Cow's milk intolerance or allergy
* Significant systemic disorder (e.g., cardiac, respiratory, endocrinological, hemato-logic, or GI); pre-pregnancy diabetes, hypertension, or other medical conditions that preclude participation per the investigator's judgement
* Taking any prescribed chronic medications
* Participation in another clinical trial
* Investigator uncertainty about the willingness or ability of the participant to comply with the protocol requirements
* Taking probiotics at screening or two weeks before enrolment
* Receiving any vaccine at screening or two weeks before enrolment

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
GI tolerance | Visit 1 (baseline, 12 weeks' gestation)
  GI tolerance via the GSRS questionnaire
GI tolerance | Visit 2 (24 weeks' gestation)
  GI tolerance via the GSRS questionnaire
GI tolerance | Visit 3 (36 weeks' gestation)
  GI tolerance via the GSRS questionnaire
GI tolerance | Visit 4 (40 days after delivery)
  GI tolerance via the GSRS questionnaire
IL-4 | Visit 1 (baseline, 12 weeks' gestation)
  Blood IL-4 levels
IL-4 | Visit 2 (24 weeks' gestation)
  Blood IL-4 levels
IL-4 | Visit 3 (36 weeks' gestation)
  Blood IL-4 levels

SECONDARY OUTCOMES:
pregnancy complications | Visit 1 (baseline, 12 weeks' gestation)
  Incidence of pregnancy complications
pregnancy complications | Visit 2 (24 weeks' gestation)
  Incidence of pregnancy complications
pregnancy complications | Visit 3 (36 weeks' gestation)
  Incidence of pregnancy complications
pregnancy complications | Visit 4 (40 days after delivery)
  Incidence of pregnancy complications
GSH levels | Visit 1 (baseline, 12 weeks' gestation)
  Blood GSH levels
GSH levels | Visit 2 (24 weeks' gestation)
  Blood GSH levels
GSH levels | Visit 3 (36 weeks' gestation)
  Blood GSH levels
IgG levels | Visit 1 (baseline, 12 weeks' gestation)
  Blood IgG levels
IgG levels | Visit 2 (24 weeks' gestation)
  Blood IgG levels
IgG levels | Visit 3 (36 weeks' gestation)
  Blood IgG levels
IL-1 levels | Visit 1 (baseline, 12 weeks' gestation)
  Blood IL-1 levels
IL-1 levels | Visit 2 (24 weeks' gestation)
  Blood IL-1 levels
IL-1 levels | Visit 3 (36 weeks' gestation)
  Blood IL-1 levels
hsCRP | Visit 1 (baseline, 12 weeks' gestation)
  Blood hsCRP levels
hsCRP | Visit 2 (24 weeks' gestation)
  Blood hsCRP levels
hsCRP | Visit 3 (36 weeks' gestation)
  Blood hsCRP levels
TNF-α | Visit 1 (baseline, 12 weeks' gestation)
  Blood TNF-α levels
TNF-α | Visit 2 (24 weeks' gestation)
  Blood TNF-α levels
TNF-α | Visit 3 (36 weeks' gestation)
  Blood TNF-α levels
Vitamin D | Visit 1 (baseline, 12 weeks' gestation)
  Blood vitamin D levels
Vitamin D | Visit 2 (24 weeks' gestation)
  Blood vitamin D levels
Vitamin D | Visit 3 (36 weeks' gestation)
  Blood vitamin D levels
Infant birth outcomes | Visit 4 (40 days after delivery)
  Infant birth outcomes, including anthropometric measurements (weight, length, head circumference, z-scores, Apgar score)
Breastmilk composition | Visit 4 (40 days after delivery)
  Breastmilk composition analyssis including metal ion testing, proteins, fats and HMOs
infant GI signs and symptoms | Visit 4 (40 days after delivery)
  infant GI signs and symptoms assessed by IGSQ questionnaire
Adverse events | Visit 1 (baseline, 12 weeks' gestation)
  Record adverse events
Adverse events | Visit 2 (24 weeks' gestation)
  Record adverse events
Adverse events | Visit 3 (36 weeks' gestation)
  Record adverse events
Adverse events | Visit 4 (40 days after delivery)
  Record adverse events

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Foshan Maternity & Child Healthcare Hospital, Foshan, Guangdong
  - Panyu Maternal and Child Care Service Centre of Guangzhou, Guangzhou, Guangdong
  - Wuxi Maternal and Child Health Hospital, Wuxi, Jiangsu
  - Affiliated hospital of Jiangnan University, Wuxi, Jiangsu
  - Xuzhou Maternal and Child Health Hospital, Xuzhou, Jiangsu
  - First People's Hospital of Chengdu, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No